CLINICAL TRIAL: NCT04819204
Title: Exploring the Role of Testosterone on Neurovascular Control in Humans
Brief Title: Testosterone and Neurovascular Control in Humans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Kevin Shoemaker, Principal Investigator, Western University, Canada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 117996
Record Dates: First submitted 2021-03-22; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GnRH antagonist alone (Experimental): Intervention: Cetrorelix acetate (Cetrotide)
  Interventions: Drug: Cetrorelix Acetate
- GnRH antagonist + Testosterone add-back (Experimental): Intervention: Cetrorelix acetate (Cetrotide) + Testosterone gel (Androgel)
  Interventions: Drug: Cetrorelix Acetate; Drug: Testosterone gel

INTERVENTIONS:
Drug: Cetrorelix Acetate — GnRH antagonist - subcutaneous injection. Day 1: 1-3 mg; Days 2-14: 0.25mg/daily.
  Other Names: Cetrotide
Drug: Testosterone gel — Testosterone gel - transdermal application of 5mg/day on Day 7-14 of GnRH antagonist
  Other Names: Androgel 1%
  Arms: GnRH antagonist + Testosterone add-back

SUMMARY:
The purpose of these studies are to evaluate the role of testosterone on autonomic and vascular function in men.

DETAILED DESCRIPTION:
Sex hormones play a pivotal role in neurovascular function in humans. In recent years, great strides have been made in elucidating the roles of estrogen and progesterone on autonomic and vascular control in women; however, very little is known about the impact of testosterone in men. Given that low testosterone levels are associated with an increased risk of cardiovascular disease, reduced exercise capacity and vascular dysfunction, it is evident that testosterone plays a pivotal role in autonomic and vascular function in men. Our current understanding of testosterone's effects on neurovascular control are confounded by numerous factors that independently alter autonomic and vascular function such as aging and chronic disease (e.g. cardiovascular disease, metabolic disease). The purpose of these studies are to evaluate the role of testosterone on autonomic and vascular function in young men to better isolate the effects of testosterone from the aforementioned confounding factors. The outcomes of these studies will provide novel information regarding the role of male sex hormones in autonomic and vascular control, and further our understanding of the influence of sex hormones on human physiology.

ELIGIBILITY:
Inclusion Criteria:

* Moderately active
* Free of chronic disease

Exclusion Criteria:

* congenital or acquired hypogonadism
* drug/alcohol dependence
* hypertension
* current smoker
* current opioid or cannabis user
* diabetes
* inability to provide written consent
* parkinson's disease
* cardiovascular disease
* testosterone use within the last year

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Muscle sympathetic nerve activity | After 7 days GnRH antagonist alone and 7 days GnRH antagonist + Testosterone
  Multi-unit postganglionic muscle sympathetic nerve activity (MSNA) will be measured by inserting a unipolar tungsten microelectrode into the peroneal nerve near the fibular head of the leg. Neural signals will be amplified, filtered (bandwidth, 700-2,000 Hz), rectified, and integrated (time constant, 0.1 s) to obtain mean voltage neurograms. MSNA will be measured during both trials to evaluate the effect of testosterone on sympathetic activity directed toward the musculature.
Endothelial function | After 7 days GnRH antagonist alone and 7 days GnRH antagonist + Testosterone
  Brachial artery flow-mediated dilation (FMD). Brachial artery FMD measures will be performed non-invasively via Doppler ultrasound.
Forearm blood flow | After 7 days GnRH antagonist alone and 7 days GnRH antagonist + Testosterone
  Forearm blood flow will be measured using Doppler ultrasound at baseline and during stress (e.g. exercise)

SECONDARY OUTCOMES:
Skeletal muscle microvascular blood flow | After 7 days GnRH antagonist alone and 7 days GnRH antagonist + Testosterone
  Microvascular blood flow will be measured using Diffuse correlation spectroscopy.

OTHER OUTCOMES:
Sex hormones | After 7 days GnRH antagonist alone and 7 days GnRH antagonist + Testosterone
  Serum concentrations of total testosterone, estradiol, albumin, and sex hormone binding globulin (SHBG) will be measured to document changes in hormone concentrations. Free testosterone will be calculated using total testosterone, SHBG and albumin.

CONTACTS AND LOCATIONS:
Overall Officials: Joel K Shoemaker, Ph.D., Principal Investigator — University of Western Ontario, Canada
Locations (1):
- the University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No